CLINICAL TRIAL: NCT04512079
Title: FREEDOM COVID Anticoagulation Strategy Randomized Trial
Brief Title: FREEDOM COVID-19 Anticoagulation Strategy
Acronym: FREEDOM COVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valentin Fuster (Other)
Responsible Party: Sponsor-Investigator, Valentin Fuster, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-2115
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Randomization; Hospitalization; PCR or Antigen Positive Test; Abnormal Laboratory Maker; Anticoagulation; Apixaban
MeSH Terms: conditions — COVID-19; Pathologic Complete Response | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized in a 1:1:1 fashion to 1 of 3 arms:
  1. Prophylactic enoxaparin (40 mg SC QD; 30 mg SC QD for CrCl <30 mL/min)
  2. Full-dose enoxaparin (1 mg/kg SC Q12h; 1 mg/kg SC QD for CrCl <30 mL/min)
  3. Apixaban (5 mg Q12h; 2.5 mg Q12h for patients with at least two of three of age ≥80 years, weight ≤60 kg or serum creatinine ≥1.5 mg/dL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prophylactic Enoxaparin (Active Comparator): Prophylactic enoxaparin (40 mg SC QD; 30 mg SC QD for CrCl <30 mL/min)
  Interventions: Drug: Enoxaparin
- Full Dose Enoxaparin (Active Comparator): Full-dose enoxaparin (1 mg/kg SC Q12h; 1 mg/kg SC QD for CrCl <30 mL/min)
  Interventions: Drug: Enoxaparin
- Apixaban (Experimental): Apixaban (5 mg Q12h; 2.5 mg Q12h for patients with at least two of three of age ≥80 years, weight ≤60 kg or serum creatinine ≥1.5 mg/dL)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Enoxaparin — Prophylactic enoxaparin (40 mg SC QD; 30 mg SC QD for CrCl <30 mL/min) Full-dose enoxaparin (1 mg/kg SC Q12h; 1 mg/kg SC QD for CrCl <30 mL/min)
  Arms: Full Dose Enoxaparin; Prophylactic Enoxaparin
Drug: Apixaban — (5 mg Q12h; 2.5 mg Q12h for patients with at least two of three of age ≥80 years, weight ≤60 kg or serum creatinine ≥1.5 mg/dL)
  Arms: Apixaban

SUMMARY:
Coronavirus Disease (COVID-19), caused by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), has led to unprecedented morbidity and mortality in the modern era. To date, nearly 13 million people have contracted COVID-19, leading to more than 550,000 deaths worldwide. As the number of affected individuals continues to climb, effective strategies for treatment and prevention of the disease are of paramount importance. SARS-CoV-2 is understood to directly invade cells via the human angiotensin-converting enzyme 2 (ACE2) receptor, which is expressed predominantly in the lungs but also throughout the cardiovascular system. Thus, while acute respiratory distress syndrome remains a feared complication, new thromboembolic disease has emerged as a common and potentially catastrophic manifestation of COVID-19.

DETAILED DESCRIPTION:
This is a Prospective, multi-center, open label, randomized controlled comparative safety and effectiveness trial with objectives: 1. To determine the effectiveness of enoxaparin and apixaban in patients hospitalized (but not yet intubated) with confirmed COVID-19 and 2. To determine the safety of enoxaparin and apixaban in patients hospitalized (but not yet intubated) with confirmed COVID-19. Observational analyses have suggested potential benefit for in-hospital use of anticoagulation. Yet, due to a lack of rigorous evidence for optimal anticoagulation regimens, practice patterns among hospitalized patients with COVID-19 vary significantly. Specifically, the choice of anticoagulant, dosing, and duration of treatment are not well understood. A preliminary analysis of approximately 2700 patients admitted to the Mount Sinai Health System (MSHS) in New York, demonstrated an association between in-hospital administration of therapeutic Anticoagulation (AC) and improved survival compared to no or prophylactic dose AC. A subsequent analysis under review of a larger 4400 patient cohort with longer follow up demonstrated similar associations with reduction in the risk of mortality and risk of intubation. Further analyses suggest more pronounced benefit with therapeutic as opposed to prophylactic doses. Bleeding rates were generally low overall, but higher among patients on therapeutic anticoagulation. Finally, though exploratory in nature, a potential signal for benefit was observed for patients on novel oral anticoagulant therapy (primarily apixaban) at therapeutic doses compared to low molecular weight heparin. Ultimately, randomized controlled trials are needed to elucidate the optimal anticoagulation regimen to improve outcomes in patients hospitalized with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization within the prior 24 hours for either confirmed (based on PCR or antigen positive test for SARS-CoV-2) or suspected COVID-19 based on 3 criteria (all 3 must be present for suspected cases):

  1. Fever >38 degrees Celsius
  2. O2 saturation ≤94
  3. Abnormal laboratory marker (at least 1):

  i. d-dimer ≥1.0 μg /mL ii. CRP >2 mg/L iii. Ferritin >300 μg /L iv. Lymphopenia <1500 cells /m3
* Patient or legal guardian provides written informed consent

Exclusion Criteria:

* Age <18 years
* Mechanical ventilation on admission or high likelihood for the need for invasive mechanical ventilation within 24 hours of admission
* Anticipated duration of hospital stay <72 hours
* Treatment with therapeutic dose UFH or LMWH, vitamin K antagonists, or NOACs within seven days
* Active bleeding
* Risk factors for bleeding, including:

  1. intracranial surgery or stroke within 3 months
  2. history of intracerebral arteriovenous malformation
  3. cerebral aneurysm or mass lesions of the central nervous system
  4. intracranial malignancy
  5. history of intracranial bleeding
  6. history of bleeding diatheses (e.g., hemophilia)
  7. history of gastrointestinal bleeding within previous 3 months
  8. thrombolysis within the previous 7 days
  9. presence of an epidural or spinal catheter
  10. recent major surgery <14 days
  11. uncontrolled hypertension (sBP > 200 mmHg or dBP > 120 mmHg)
  12. other physician-perceived contraindications to anticoagulation
  13. Platelet count <50 x109/L, INR >2.0, or baseline aPTT >50 seconds
  14. Hemoglobin <80 g/L (to minimize the likelihood of requiring red blood cell transfusion if potential bleeding were to occur)
  15. current treatment with antithrombotics or antiplatelet agents including but not limited to ticagrelor, prasugrel, and aspirin> 100mg, or non-steroidal anti-inflammatory drugs (e.g. ibuprofen, naproxen, etc.) due to increased risk of bleeding, unless such agents can be permanently discontinued (aspirin <= 100mg and clopidogrel <=75mg is permitted)
* Acute or subacute bacterial endocarditis
* History of heparin induced thrombocytopenia (HIT) or other heparin allergy including hypersensitivity
* Patients with non-COVID-19 related clinical condition for which life expectancy is <6 months
* Pregnancy (women of childbearing potential are required to have a negative pregnancy test prior to enrollment)
* Active enrollment in other trials related to anticoagulation
* Patients has end stage kidney disease (ESKD) on chronic dialysis
* Patient is a member of a vulnerable population: In the judgment of the investigator the patient is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3460 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Time to first event | 30 days
  The time to first event rate within 30 days of randomization of the composite of all-cause mortality, intubation requiring mechanical ventilation, systemic thromboembolism (including pulmonary emboli) confirmed by imaging or requiring surgical intervention OR ischemic stroke confirmed by imaging.
Number of in-hospital rate of BARC 3 or 5 | 30 days
  Number of in-hospital rate of BARC 3 or 5 bleeding (binary). BARC Type 3: a. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  b. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  c. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision. BARC Type 5:
  1. Probable fatal bleeding
  2. Definite fatal bleeding (overt or autopsy or imaging confirmation)

SECONDARY OUTCOMES:
Number of participants with Myocardial infarction | 30 days after randomization
  Myocardial infarction (according to the 4th universal definition, types 1,2, and 3)
Number of participants with Myocardial infarction | 90 days after randomization
  Myocardial infarction (according to the 4th universal definition, types 1,2, and 3)
Number of participants with Deep Vein Thrombosis | 30 days after randomization
  Deep vein thrombosis with confirmation on imaging
Number of participants with Deep Vein Thrombosis | 90 days after randomization
  Deep vein thrombosis with confirmation on imaging
Number of participants requiring Ventilation | 30 after randomization
  Intubation and mechanical ventilation
Number of participants requiring Ventilation | 90 days after randomization
  Intubation and mechanical ventilation
Number of All Death | 30 days after randomization
  All-cause death
Number of All Death | 90 days after randomization
  All-cause death
Cause of Death | 30 days after randomization
  Cause of Death
Cause of Death | 90 days after randomization
  Cause of Death
Number of participants with Stroke | 30 days after randomization
  Stroke confirmed by imaging or autopsy (all, ischemic and hemorrhagic)
Number of participants with Stroke | 90 days after randomization
  Stroke confirmed by imaging or autopsy (all, ischemic and hemorrhagic)
Number of participants with Pulmonary Emboli | 30 days after randomization
  Pulmonary emboli confirmed by imaging or autopsy
Number of participants with Pulmonary Emboli | 90 days after randomization
  Pulmonary emboli confirmed by imaging or autopsy
Number of participants with Systemic Thromboembolism | 30 days after randomization
  Systemic thromboembolism confirmed by imaging or requiring surgical intervention
Number of participants with Systemic Thromboembolism | 90 days after randomization
  Systemic thromboembolism confirmed by imaging or requiring surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD,PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Anu Lala, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (21):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Brazil (2):
  - Instituto do Coração - INCOR, São Paulo
  - Instituto Prevent Senior - IPS, São Paulo
- Colombia (6):
  - Clínica de la Costa, Barranquilla
  - Clínica Shaio, Bogotá
  - Fundación Cardioinfantil, Bogotá
  - Fundacion Oftalmológica de Santander - Foscal, Bucaramanga
  - Centro Médico Imbanaco, Cali
  - CardioVid, Medellín
- India (7):
  - Eternal Heart Care Centre and Research Ins Pvt Ltd., Jaipur
  - Jaipur National University, Jaipur
  - Sawai Mann Singh Hospital, Jaipur
  - Jaslok Hospital & Research Center, Mumbai
  - Saifee Hospital, Mumbai
  - Sengupta Hospital & Research Institute, Nagpur
  - D Y Patil University School of Medicine & D Y Patil Hospital, Navi Mumbai
- Mexico (5):
  - Hospital Cardiológica Aguascalientes, Aguascalientes
  - Centro Médico Nacional 20 de Noviembre, Mexico City
  - Christus Muguerza Hospital Alta Especialidad, Monterrey
  - Centro de Estudios Clinicos de Querétaro S.C., Querétaro City
  - Centro Medico Hospital del Prado, Tijuana

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. The type of analysis that will be conducted is for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Derived] Stone GW, Farkouh ME, Lala A, Tinuoye E, Dressler O, Moreno PR, Palacios IF, Goodman SG, Esper RB, Abizaid A, Varade D, Betancur JF, Ricalde A, Payro G, Castellano JM, Hung IFN, Nadkarni GN, Giustino G, Godoy LC, Feinman J, Camaj A, Bienstock SW, Furtado RHM, Granada C, Bustamante J, Peyra C, Contreras J, Owen R, Bhatt DL, Pocock SJ, Fuster V; FREEDOM COVID Anticoagulation Strategy Randomized Trial Investigators. Randomized Trial of Anticoagulation Strategies for Noncritically Ill Patients Hospitalized With COVID-19. J Am Coll Cardiol. 2023 May 9;81(18):1747-1762. doi: 10.1016/j.jacc.2023.02.041. Epub 2023 Mar 6. PMID 36889611
- [Derived] Farkouh ME, Stone GW, Lala A, Bagiella E, Moreno PR, Nadkarni GN, Ben-Yehuda O, Granada JF, Dressler O, Tinuoye EO, Granada C, Bustamante J, Peyra C, Godoy LC, Palacios IF, Fuster V. Anticoagulation in Patients With COVID-19: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Mar 8;79(9):917-928. doi: 10.1016/j.jacc.2021.12.023. PMID 35241226